CLINICAL TRIAL: NCT01712009
Title: Randomized, Phase 2 Study to Estimate the Effect of Prophylactic Intervention With Naproxen or Loratadine on Bone Pain in Breast Cancer Subjects Receiving Chemotherapy and Pegfilgrastim
Brief Title: NOLAN: Naproxen or Loratadine and Neulasta
Acronym: NOLAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110147
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Bone Pain in Stage I - III Breast Cancer
Keywords: Breast cancer; Chemotherapy; Neulasta; Pegfilgrastim; Naproxen; Loratadine; Non-steroidal antiinflammatory drug (NSAID); Anti-histamine; Bone Pain
MeSH Terms: conditions — Breast Neoplasms | interventions — Naproxen; Loratadine; pegfilgrastim; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prophylactic naproxen (Experimental): Participants received adjuvant or neoadjuvant chemotherapy with pegfilgrastim prophylaxis in addition to prophylactic naproxen 500 mg orally twice a day (BID) for 5 days in each of the 4 cycles, beginning on the day of pegfilgrastim administration.
  Interventions: Drug: Naproxen; Biological: Pegfilgrastim; Drug: Chemotherapy
- Prophylactic loratadine (Experimental): Participants received adjuvant or neoadjuvant chemotherapy with pegfilgrastim prophylaxis in addition to prophylactic loratadine 10 mg once a day (QD) for 5 days in each of the 4 cycles, beginning on the day of pegfilgrastim administration.
  Interventions: Drug: Loratadine; Biological: Pegfilgrastim; Drug: Chemotherapy
- No prophylactic treatment (Other): Participants received adjuvant or neoadjuvant chemotherapy with pegfilgrastim prophylaxis.
  Interventions: Biological: Pegfilgrastim; Drug: Chemotherapy

INTERVENTIONS:
Drug: Naproxen
  Arms: Prophylactic naproxen
Drug: Loratadine
  Arms: Prophylactic loratadine
Biological: Pegfilgrastim — Commercially available pegfilgrastim (Neulasta®) will be used in the study, and is considered background therapy. Pegfilgrastim is administered as a single 6 mg subcutaneous injection 24 hours to 72 hours after completion of chemotherapy.
  Other Names: Neulasta®
Drug: Chemotherapy — The choice of chemotherapy regimen (agent, dose, and schedule) is at the discretion of the treating physician.

SUMMARY:
The primary objective of the study is to estimate the difference in bone pain between breast cancer patients receiving chemotherapy and pegfilgrastim and either no prophylactic intervention, prophylactic naproxen, or prophylactic loratadine.

DETAILED DESCRIPTION:
In this study, the investigational products are naproxen, a non-steroidal antiinflammatory drug (NSAID), and loratadine, an anti-histamine. Both agents are being investigated as prophylactic medications to reduce the incidence and/or severity of bone pain in breast cancer patients receiving adjuvant or neoadjuvant myelosuppressive chemotherapy and pegfilgrastim prophylaxis.

Pegfilgrastim treatment is used to stimulate bone marrow to produce more neutrophils to help fight infections in patients undergoing chemotherapy.

ELIGIBILITY:
Age 18 years or over

* Eastern cooperative oncology group (ECOG) performance status 0-2
* Female with newly diagnosed, not previously treated with chemotherapy, stage I-III breast cancer
* Medically eligible to safely receive adjuvant or neoadjuvant chemotherapy, pegfilgrastim, naproxen and loratadine as determined by the investigator
* Creatinine ≤ 1.5 X upper limit of normal (ULN)
* Planning to receive at least 4 cycles of adjuvant or neoadjuvant chemotherapy
* Planning to receive prophylaxis with pegfilgrastim starting in the first cycle and continuing throughout each chemotherapy cycle of the treatment period
* Subject has provided informed consent

Exclusion Criteria

* History of other malignancy within the past 5 years, with the following exceptions:

  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Planning to receive weekly chemotherapy
* Ongoing chronic pain, or other painful conditions requiring treatment (including immediate post-operative treatment of surgical or procedural-associated pain) as determined by the investigator
* Chronic oral steroid use. Premedication related to the administration of chemotherapy, and use of anti-emetics is allowed, per usual clinical practice
* Chronic use of oral non-steroidal anti-inflammatory drug (NSAIDs) or oral antihistamines outside of those dictated by the randomization groups outlined in the protocol, with the following exception:

  - Chronic oral aspirin use for cardiovascular-related indications
* Prior chemotherapy treatment for cancer within 5 years of current breast cancer diagnosis
* Prior use of granulocyte colony stimulating factor (G-CSF)
* History of clinically significant gastrointestinal (GI) bleeding, history of GI ulcers or active GI bleeding within 6 months prior to randomization
* History of clinically significant bleeding disorders, thromboembolism within 6 months prior to randomization
* Currently enrolled in, or less than 30 days since ending, another clinical trial which includes language directing G-CSF (filgrastim, pegfilgrastim, other) or granulocyte-macrophage colony-stimulating factor (GM-CSF) (sargramostim) use
* Currently enrolled in, or less than 30 days since ending, another interventional clinical trial which includes a blinded treatment or blinded treatment arm (whether or not the subject is randomized to the blinded arm)
* Currently enrolled in, or less than 30 days since ending, another interventional clinical trial which includes the use of any agent not currently considered to be standard therapy for the adjuvant or neoadjuvant treatment of stage I-III breast cancer based on National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology for Breast Cancer
* Currently enrolled in, or less than 30 days since ending, any pain intervention study
* Female subjects who are pregnant or lactating or of reproductive potential not willing to employ an effective method of birth control during treatment and for 17 days after discontinuing study treatment
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the Investigator or Amgen, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2015-03-18 (Actual); Study Completion 2015-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (81):
- United States (81):
  - Research Site, Muscle Shoals, Alabama
  - Research Site, Anaheim, California
  - Research Site, Fullerton, California
  - Research Site, Santa Maria, California
  - Research Site, Santa Rosa, California
  - Research Site, Torrance, California
  - Research Site, Whittier, California
  - Research Site, Denver, Colorado
  - Research Site, Golden, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Norwich, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Lakeland, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Plantation, Florida
  - Research Site, Stuart, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Thomasville, Georgia
  - Research Site, Elmhurst, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Mount Vernon, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Sioux City, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Hutchinson, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Mount Sterling, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Marrero, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Cumberland, Maryland
  - Research Site, Randallstown, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Westminster, Maryland
  - Research Site, Lowell, Massachusetts
  - Research Site, Battle Creek, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Saint Joseph, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Nashua, New Hampshire
  - Research Site, Denville, New Jersey
  - Research Site, East Syracuse, New York
  - Research Site, Johnson City, New York
  - Research Site, Gastonia, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Massillon, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Bend, Oregon
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Florence, South Carolina
  - Research Site, Watertown, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Chattanooga, Tennessee
  - Research Site, Corpus Christi, Texas
  - Research Site, Plano, Texas
  - Research Site, Ogden, Utah
  - Research Site, Chesapeake, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Huntington, West Virginia
  - Research Site, Janesville, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Racine, Wisconsin
  - Research Site, Wauwatosa, Wisconsin
  - Research Site, Weston, Wisconsin

REFERENCES:
- [Background] Kirshner JJ, McDonald MC 3rd, Kruter F, Guinigundo AS, Vanni L, Maxwell CL, Reiner M, Upchurch TE, Garcia J, Morrow PK. NOLAN: a randomized, phase 2 study to estimate the effect of prophylactic naproxen or loratadine vs no prophylactic treatment on bone pain in patients with early-stage breast cancer receiving chemotherapy and pegfilgrastim. Support Care Cancer. 2018 Apr;26(4):1323-1334. doi: 10.1007/s00520-017-3959-2. Epub 2017 Nov 16. PMID 29147854
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 83 centers in the United States. The first participant enrolled on 01 November 2012 and the last participant enrolled on 20 November 2014.
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to receive no prophylactic intervention, prophylactic naproxen, or prophylactic loratadine. Randomization was stratified by age group (< 65 years vs ≥ 65 years) and planned chemotherapy type (taxane vs non-taxane). Participants remained on study for the first 4 chemotherapy cycles.
Groups:
- No Prophylaxis: Participants received adjuvant or neoadjuvant chemotherapy and pegfilgrastim.
- Naproxen 500 mg BID: Participants received adjuvant or neoadjuvant chemotherapy and pegfilgrastim in addition to prophylactic naproxen 500 mg orally twice a day (BID) for 5 days in each of the 4 cycles, beginning on the day of pegfilgrastim administration.
- Loratadine 10 mg QD: Participants received adjuvant or neoadjuvant chemotherapy and pegfilgrastim in addition to prophylactic loratadine 10 mg once a day (QD) for 5 days in each of the 4 cycles, beginning on the day of pegfilgrastim administration.
Period: Overall Study
Arm/Group | No Prophylaxis | Naproxen 500 mg BID | Loratadine 10 mg QD
Started | 198 | 200 | 202
Received Pegfilgrastim | 191 | 196 | 200
Received Naproxen / Loratadine | 0 | 193 | 198
Completed | 160 | 171 | 181
Not Completed | 38 | 29 | 21
Not completed — Withdrawal by Subject | 24 | 15 | 8
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Decision by Sponsor | 12 | 14 | 12

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants based on the randomization treatment group who received primary prophylaxis with pegfilgrastim.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Prophylaxis | Naproxen 500 mg BID | Loratadine 10 mg QD | Total
Number analyzed (Participants) | 191 | 196 | 200 | 587
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.7) | 53.2 (11.7) | 54.6 (10.9) | 54.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 196 | 200 | 587
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 13 | 15 | 9 | 37
  Not Hispanic/Latino | 178 | 181 | 191 | 550
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 3 | 1 | 7
  Black (or African American) | 33 | 27 | 23 | 83
  Multiple | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  White | 148 | 166 | 173 | 487
  Other | 5 | 0 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Bone Pain (All Grades) in Cycle 1
Description: Bone pain data were captured as part of standard adverse event (AE) reporting.
Time Frame: Cycle 1 (approximately 4 weeks, depending on the chemotherapy dosing interval)
Population: Full anlysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No Prophylaxis | Naproxen 500 mg BID | Loratadine 10 mg QD
Number analyzed (Participants) | 191 | 196 | 200
percentage of participants | 46.6 [39.4 to 53.9] | 40.3 [33.4 to 47.5] | 42.5 [35.6 to 49.7]
Statistical Analysis 1: Comparison: No Prophylaxis vs Naproxen 500 mg BID; Test type: Superiority or Other; Difference = -6.3, 95% CI 2-sided [-16.7 to 4.1] — Naproxen minus No Prophylaxis
Statistical Analysis 2: Comparison: No Prophylaxis vs Loratadine 10 mg QD; Test type: Superiority or Other; Difference = -4.1, 95% CI 2-sided [-14.5 to 6.3] — Loratadine minus No Prophylaxis
Statistical Analysis 3: Comparison: Naproxen 500 mg BID vs Loratadine 10 mg QD; Test type: Superiority or Other; Difference = 2.2, 95% CI 2-sided [-8.0 to 12.4] — Loratadine minus Naproxen

2. Secondary Outcome: Percentage of Participants With Bone Pain (All Grades) by Cycle (2-4) and Across Cycles
Description: Bone pain data were captured as part of standard adverse event (AE) reporting.
Time Frame: Cycles 1, 2, 3 and 4 (approximately 4 weeks each, depending on the chemotherapy dosing interval)
Population: Full analysis set; "n" indicates the number of participants who entered each cycle.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No Prophylaxis | Naproxen 500 mg BID | Loratadine 10 mg QD
Number analyzed (Participants) | 191 | 196 | 200
percentage of participants
  Cycle 2 (n=178, 180, 193) | 34.3 [27.3 to 41.7] | 34.4 [27.5 to 41.9] | 34.7 [28.0 to 41.9]
  Cycle 3 (n=165, 176, 188) | 33.9 [26.8 to 41.7] | 34.1 [27.1 to 41.6] | 36.2 [29.3 to 43.5]
  Cycle 4 (n=162, 169, 179) | 40.7 [33.1 to 48.7] | 40.2 [32.8 to 48.0] | 38.0 [30.9 to 45.5]
  Across All Cycles (n=191, 196, 200) | 63.4 [56.1 to 70.2] | 59.2 [52.0 to 66.1] | 61.0 [53.9 to 67.8]
Statistical Analysis 1: Comparison: No Prophylaxis vs Naproxen 500 mg BID; Difference across all treatment cycles; Test type: Superiority or Other; Difference = -4.2, 95% CI 2-sided [-14.4 to 6.0] — Naproxen minus No Prophylaxis
Statistical Analysis 2: Comparison: No Prophylaxis vs Loratadine 10 mg QD; Difference across all treatment cyces; Test type: Superiority or Other; Difference = -2.4, 95% CI 2-sided [-12.5 to 7.8] — Loratadine minus No Prophylaxis
Statistical Analysis 3: Comparison: Naproxen 500 mg BID vs Loratadine 10 mg QD; Dfference across all treatment cycles; Test type: Superiority or Other; Difference = 1.8, 95% CI 2-sided [-8.3 to 12.0] — Loratadine minus Naproxen

3. Secondary Outcome: Percentage of Participants With Severe Bone Pain by Cycle and Across Cycles
Description: Bone pain data were captured as part of standard adverse event reporting. Severe bone pain is defined as grade 3 or 4 according to common terminology criteria for adverse events (CTCAE) version 3 grading criteria: Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, and Grade 4 = Life-threatening or disabling.
Time Frame: Cycles 1, 2, 3 and 4 (approximately 4 weeks each, depending on the chemotherapy dosing interval)
Population: Full analysis set; "n" indicates the number of participants who entered each cycle.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No Prophylaxis | Naproxen 500 mg BID | Loratadine 10 mg QD
Number analyzed (Participants) | 191 | 196 | 200
percentage of participants
  Cycle 1 (n=191, 196, 200) | 4.7 [2.2 to 8.8] | 3.1 [1.1 to 6.5] | 4.5 [2.1 to 8.4]
  Cycle 2 (n=178, 180, 193) | 1.1 [0.1 to 4.0] | 1.7 [0.3 to 4.8] | 0.0 [0.0 to 1.9]
  Cycle 3 (n=165, 176, 188) | 1.8 [0.4 to 5.2] | 1.1 [0.1 to 4.0] | 0.0 [0.0 to 1.9]
  Cycle 4 (n=162, 169, 179) | 1.9 [0.4 to 5.3] | 0.6 [0.0 to 3.3] | 0.0 [0.0 to 2.0]
  Across All Cycles (n=191, 196, 200) | 5.8 [2.9 to 10.1] | 4.1 [1.8 to 7.9] | 4.5 [2.1 to 8.4]
Statistical Analysis 1: Comparison: No Prophylaxis vs Naproxen 500 mg BID; Difference across all treatment cycles; Test type: Superiority or Other; Difference = -1.7, 95% CI 2-sided [-6.5 to 3.2] — Naproxen minus No Prophylaxis
Statistical Analysis 2: Comparison: No Prophylaxis vs Loratadine 10 mg QD; Difference across all cycles; Test type: Superiority or Other; Difference = -1.3, 95% CI 2-sided [-6.1 to 3.6] — Loratadine minus No Prophylaxis
Statistical Analysis 3: Comparison: Naproxen 500 mg BID vs Loratadine 10 mg QD; Difference across all cycles; Test type: Superiority or Other; Difference = 0.4, 95% CI 2-sided [-4.1 to 4.9] — Loratadine minus Naproxen

4. Secondary Outcome: Mean Patient-reported Bone Pain by Cycle and Across Cycles
Description: Participants completed a brief bone pain survey once per day for 5 days beginning the day they received their pegfilgrastim injection. The bone pain survey collected the severity of pain using a 0 (no pain) to 10 (worst pain) scale. Mean patient-reported bone pain values are the average of each participant's bone pain values across survey days 1-5 within each cycle. Across all cycles the mean is the average of each patient-reported bone pain value across all survey days 1-5 and across all cycles. An analysis of variance (ANOVA) model with treatment as explanatory term was used.
Time Frame: Five consecutive days during each cycle beginning on the day of pegfilgrastim administration (Day 2, 3, or 4 of each cycle)
Population: Full analysis set; all missing values of patient-reported bone pain within any cycle were imputed. "n" indicates the number of participants who entered each cycle.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | No Prophylaxis | Naproxen 500 mg BID | Loratadine 10 mg QD
Number analyzed (Participants) | 191 | 196 | 200
units on a scale
  Cycle 1 (n=191, 196, 200) | 2.2 (0.2) | 1.8 (0.2) | 1.7 (0.1)
  Cycle 2 (n=178, 180, 193) | 1.7 (0.2) | 1.3 (0.1) | 1.4 (0.1)
  Cycle 3 (n=165, 176, 188) | 1.6 (0.2) | 1.3 (0.1) | 1.4 (0.1)
  Cycle 4 (n=162, 169, 179) | 1.7 (0.2) | 1.2 (0.1) | 1.3 (0.1)
  Across all Cycles (n=191, 196, 200) | 1.9 (0.1) | 1.5 (0.1) | 1.5 (0.1)
Statistical Analysis 1: Comparison: No Prophylaxis vs Naproxen 500 mg BID; Difference across all treatment cycles; Test type: Superiority or Other; p = 0.0881, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.7 to 0.0], Standard Error of Mean 0.2 — Naproxen minus No Prophylaxis
Statistical Analysis 2: Comparison: No Prophylaxis vs Loratadine 10 mg QD; Difference across all treatment cycles; Test type: Superiority or Other; p = 0.0443, ANOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.0], Standard Deviation 0.2 — Loratadine minus No Prophylaxis
Statistical Analysis 3: Comparison: Naproxen 500 mg BID vs Loratadine 10 mg QD; Difference across all treatment cycles; Test type: Superiority or Other; p = 0.8007, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.4 to 0.3], Standard Error of Mean 0.2 — Loratadine minus Naproxen

5. Secondary Outcome: Maximum Patient-reported Bone Pain by Cycle and Across Cycles
Description: Participants completed a brief bone pain survey once per day for 5 days beginning the day they received their pegfilgrastim injection. The bone pain survey collected the severity of pain using a 0 (no pain) to 10 (worst pain) scale. Maximum patient-reported bone pain is the maximum of each participant's bone pain values across survey Days 1-5 within each cycle. Across all cycles the maximum is the maximum of each patient-reported bone pain value across all survey days 1-5 and across all cycles. An ANOVA model with treatment as explanatory term was used.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | No Prophylaxis | Naproxen 500 mg BID | Loratadine 10 mg QD
Number analyzed (Participants) | 191 | 196 | 200
units on a scale
  Cycle 1 (n=191, 196, 200) | 3.9 (0.2) | 3.3 (0.2) | 3.0 (0.2)
  Cycle 2 (n=178, 180, 193) | 3.0 (0.2) | 2.4 (0.2) | 2.6 (0.2)
  Cycle 3 (n=165, 176, 188) | 2.7 (0.2) | 2.2 (0.2) | 2.5 (0.2)
  Cycle 4 (n=162, 169, 179) | 2.8 (0.2) | 2.1 (0.2) | 2.1 (0.2)
  Across All Cycles (n=191, 196, 200) | 4.7 (0.2) | 4.2 (0.2) | 4.1 (0.2)
Statistical Analysis 1: Comparison: No Prophylaxis vs Naproxen 500 mg BID; Difference across all treatment cycles; Test type: Superiority or Other; p = 0.1466, ANOVA; LS Mean Difference = -0.5, 95% CI 2-sided [-1.1 to 0.2], Standard Error of Mean 0.3 — Naproxen minus No Prophylaxis
Statistical Analysis 2: Comparison: No Prophylaxis vs Loratadine 10 mg QD; Difference across all treatment cycles; Test type: Superiority or Other; p = 0.0411, ANOVA; LS Mean Difference = -0.7, 95% CI 2-sided [-1.3 to -0.0], Standard Error of Mean 0.3 — Loratadine minus No Prophylaxis
Statistical Analysis 3: Comparison: Naproxen 500 mg BID vs Loratadine 10 mg QD; Difference across all treatment cycles; Test type: Superiority or Other; p = 0.5689, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.8 to 0.5], Standard Error of Mean 0.3 — Loratadine minus Naproxen

6. Secondary Outcome: Area Under the Curve (AUC) for Patient-reported Bone Pain
Description: Patient-reported bone pain AUC was calculated using the trapezoidal rule with bone pain scores from day 1 to 5 for each cycle. The AUC across cycles is the average of AUCs across the cycle.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale * days
Arm/Group | No Prophylaxis | Naproxen 500 mg BID | Loratadine 10 mg QD
Number analyzed (Participants) | 191 | 196 | 200
units on a scale * days
  Cycle 1 (n=191, 196, 200) | 9.3 (0.7) | 7.7 (0.6) | 7.0 (0.6)
  Cycle 2 (n=178, 180, 193) | 7.3 (0.7) | 5.6 (0.6) | 5.9 (0.5)
  Cycle 3 (n=165, 176, 188) | 6.8 (0.7) | 5.5 (0.6) | 6.1 (0.6)
  Cycle 4 (n=162, 169, 179) | 7.2 (0.7) | 5.2 (0.6) | 5.6 (0.6)
  Across All Cycles (n=191, 196, 200) | 8.0 (0.6) | 6.6 (0.5) | 6.3 (0.5)
Statistical Analysis 1: Comparison: No Prophylaxis vs Naproxen 500 mg BID; Difference across all treatment cycles; Test type: Superiority or Other; p = 0.0775, ANOVA; LS Mean Difference = -1.4, 95% CI [-3.0 to 0.2], Standard Error of Mean 0.8 — Naproxen minus No Prophylaxis
Statistical Analysis 2: Comparison: No Prophylaxis vs Loratadine 10 mg QD; Difference across all treatment cycles; Test type: Superiority or Other; p = 0.0329, ANCOVA; LS Mean Difference = -1.6, 95% CI 2-sided [-3.1 to -0.1], Standard Error of Mean 0.8 — Loratadine minus No Prophylaxis
Statistical Analysis 3: Comparison: Naproxen 500 mg BID vs Loratadine 10 mg QD; Difference across all treatment groups; Test type: Superiority or Other; p = 0.7572, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-1.7 to 1.2], Standard Error of Mean 0.7 — Loratadine minus Naproxen

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Severity was graded using CTCAE version 3. A serious adverse event (SAE) is defined as an adverse event that meets at least 1 of the following serious criteria: • fatal; • life threatening; • requires in-patient hospitalization or prolongation of existing hospitalization; • results in persistent or significant disability/incapacity; • congenital anomaly/birth defect; • other medically important serious event.
  The investigator assessed each adverse event for relatedness to investigational product(s) or other protocol-required therapies.
Time Frame: From first dose of investigational product (IP, naproxen or loratidine) or first dose of pegfilgrastim (Peg), whichever occurred first, until 30 days after last dose, up to 24 weeks.
Population: Safety analysis set included all participants who received primary prophylaxis with pegfilgrastim according to the prophylactic medication actually received. Participants in the Naproxen or Loratadine groups who did not receive naproxen or loratadine are analyzed in the No Prophylaxis group for safety analyses.
Measure: Number; unit: participants
Arm/Group | No Prophylaxis | Naproxen 500 mg BID | Loratadine 10 mg QD
Number analyzed (Participants) | 196 | 193 | 198
participants
  Any adverse event | 188 | 192 | 194
  Worst grade of ≥ 2 | 164 | 169 | 168
  Worst grade of ≥ 3 | 74 | 73 | 63
  Worst grade of ≥ 4 | 18 | 30 | 20
  Serious adverse events | 34 | 30 | 14
  Fatal adverse events | 0 | 0 | 0
  AE leading to discontinuation from study | 3 | 5 | 3
  SAE leading to discontinuation from study | 1 | 3 | 2
  Any adverse event related to IP | 0 | 30 | 7
  SAE related to IP | 0 | 1 | 0
  AE related to IP leading to discontinuation of IP | 0 | 9 | 0
  SAE related to IP leading to discontinuation of IP | 0 | 1 | 0
  Any adverse event related to pegfilgrastim | 87 | 96 | 105
  SAE related to pegfilgrastim | 4 | 0 | 1
  AE related to / leading to discontinuation of Peg | 6 | 3 | 6
  SAE related to / leading to discontinuation of Peg | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of investigational product (naproxen or loratidine) or first dose of pegfilgrastim, whichever occurred first, until 30 days after last dose, up to 24 weeks.
Description: Participants in the Naproxen or Loratadine groups who did not receive naproxen or loratadine are analyzed in the No Prophylaxis group for safety analyses.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- No Prophylactic Intervention: Participants received adjuvant or neoadjuvant chemotherapy and pegfilgrastim.
- Naproxen 500mg BID: Participants received adjuvant or neoadjuvant chemotherapy and pegfilgrastim in addition to prophylactic naproxen 500 mg orally twice a day (BID) for 5 days in each of the 4 cycles, beginning on the day of pegfilgrastim administration.
- Loratadine 10mg QD: Participants received adjuvant or neoadjuvant chemotherapy and pegfilgrastim in addition to prophylactic loratadine 10 mg once a day (QD) for 5 days in each of the 4 cycles, beginning on the day of pegfilgrastim administration.
Arm/Group | No Prophylactic Intervention | Naproxen 500mg BID | Loratadine 10mg QD
Serious Adverse Events (participants affected / at risk) | 34/196 | 30/193 | 14/198
Other Adverse Events (participants affected / at risk) | 184/196 | 190/193 | 193/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Prophylactic Intervention (N=196) | Naproxen 500mg BID (N=193) | Loratadine 10mg QD (N=198)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 6 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Abscess bacterial (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Fungaemia (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Implant site abscess (Infections and infestations) | 0 | 1 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 2 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incorrect drug administration duration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 3 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 4 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No Prophylactic Intervention (N=196) | Naproxen 500mg BID (N=193) | Loratadine 10mg QD (N=198)
Anaemia (Blood and lymphatic system disorders) | 42 | 60 | 40
Leukopenia (Blood and lymphatic system disorders) | 10 | 10 | 7
Lymphopenia (Blood and lymphatic system disorders) | 2 | 10 | 2
Neutropenia (Blood and lymphatic system disorders) | 19 | 27 | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 15 | 9
Lacrimation increased (Eye disorders) | 5 | 5 | 15
Abdominal pain (Gastrointestinal disorders) | 14 | 11 | 5
Constipation (Gastrointestinal disorders) | 60 | 77 | 66
Diarrhoea (Gastrointestinal disorders) | 67 | 75 | 71
Dyspepsia (Gastrointestinal disorders) | 26 | 29 | 25
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 | 16 | 12
Nausea (Gastrointestinal disorders) | 98 | 118 | 100
Stomatitis (Gastrointestinal disorders) | 30 | 32 | 38
Vomiting (Gastrointestinal disorders) | 32 | 43 | 29
Asthenia (General disorders) | 10 | 8 | 9
Fatigue (General disorders) | 120 | 110 | 128
Mucosal inflammation (General disorders) | 18 | 21 | 23
Oedema peripheral (General disorders) | 18 | 17 | 19
Pain (General disorders) | 23 | 17 | 22
Pyrexia (General disorders) | 14 | 18 | 15
Upper respiratory tract infection (Infections and infestations) | 11 | 8 | 6
Urinary tract infection (Infections and infestations) | 9 | 12 | 3
Neutrophil count decreased (Investigations) | 7 | 4 | 10
White blood cell count decreased (Investigations) | 13 | 6 | 10
Decreased appetite (Metabolism and nutrition disorders) | 36 | 34 | 39
Dehydration (Metabolism and nutrition disorders) | 20 | 14 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 10 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 17 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 31 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 16 | 17
Bone pain (Musculoskeletal and connective tissue disorders) | 56 | 55 | 63
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 18 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 17 | 22
Dizziness (Nervous system disorders) | 26 | 15 | 15
Dysgeusia (Nervous system disorders) | 14 | 20 | 32
Headache (Nervous system disorders) | 49 | 54 | 48
Neuropathy peripheral (Nervous system disorders) | 14 | 24 | 24
Paraesthesia (Nervous system disorders) | 7 | 3 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 11 | 6
Anxiety (Psychiatric disorders) | 16 | 20 | 11
Depression (Psychiatric disorders) | 11 | 6 | 7
Insomnia (Psychiatric disorders) | 22 | 35 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 25 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 17 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 17
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 13 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 68 | 85 | 106
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 8 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 9 | 9
Rash (Skin and subcutaneous tissue disorders) | 23 | 23 | 29
Hot flush (Vascular disorders) | 16 | 12 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.